CLINICAL TRIAL: NCT02401074
Title: Role of Airway Tissue Temperature in Asthma Exacerbation
Brief Title: Airway Temperature
Acronym: RATE
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was withdrawn prior to patient enrollment due to COVID-19, funding termination and lack of eligible study participants.
Sponsor: Lu Yuan Lee (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Lu Yuan Lee, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IND 16362; U01AI123832 (NIH)
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Allergens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Segmental bronchoprovocation with Allergen (SBP-Ag) (Experimental): Following nasopharyngeal anesthesia, the fiberoptic bronchoscope will then be passed into a pulmonary segment or subsegment. During SBP-Ag challenge, 15% of the Ag-PD20 allergenic extract will be instilled into the segment.
  Interventions: Biological: Segmental Bronchoprovocation with Allergen (SBP-Ag)

INTERVENTIONS:
Biological: Segmental Bronchoprovocation with Allergen (SBP-Ag) — Premedication will consist of intramuscular glycopyrolate (0.2 mg), and midazolam (0.5-2.0 mg). Subjects will also be given a short-acting beta agonist, albuterol (2 puffs, 180 mcg) prior to bronchoscopy. Following nasopharyngeal anesthesia (topical lidocaine), the fiberoptic bronchoscope will then be passed into a pulmonary segment or subsegment. During the SBP-Ag challenge, approximately 15% of the Ag-PD20 allergenic extract will be instilled into the segment (5)

SUMMARY:
Airway irritation, cough and bronchial spasm are common symptoms in patients with airway inflammatory diseases such as asthma. The primary focus of this exploratory study is to determine if there is an increase in tissue temperature in airway mucosa during asthma exacerbation. The results of this study will bring a better understanding of the potential involvement of an increase in airway mucosa temperature in the pathogenesis of various symptoms in these patients. The finding should help to advance the development of new therapeutic strategies for these debilitating diseases.

DETAILED DESCRIPTION:
A total of eight participants will be enrolled into this study. We will take direct measurements of bronchial mucosa temperature. This can only be tested accurately in asthma participants because anesthesia is known to lower the body temperature. The proposed study using and experimental procedure called a segmental bronchoprovocation challenge with allergen in asthmatic patients offers a unique approach to test our hypothesis.

Individuals enrolled into this study will participate for eight weeks and will take part in four visits each estimated to last 2 and 8 hours. Participants will also participant in one follow-up phone call following Test day 2.

Patients with asthma and healthy participants will be recruited to participate in this study through advertisement postings in the Kentucky Clinic and/or the University of Kentucky Hospital as well as on main campus. The study will also be added to a website using the same posting.

Patients with asthma who have been prescribed for a diagnostic or therapeutic bronchoscopy procedure at the UK Pulmonary Clinic will be identified and recruited by qualified physicians in that clinic. The medical history and records of the patients will be made available which includes data form a complete spirometry test and other clinical tests, physical examination, smoking history, symptoms, current medication use, drug allergies, laboratory and imaging data.

After eligible patients are identified and meet proper inclusion criteria, informed consent will be obtained.

Participants will receive an explanation of the research project including any potential risks. In addition, the participant will be shown the actual size of the temperature probe to be used in this procedure. The participation of these individuals in the study will in no way affect their current treatment. No bias will be held against the individual by any clinical staff if they elect not to participate in the study. Informed consent will be obtained after the potential participant is fully informed via verbal/written information of the procedures and nature of the research, the risks involved, and their rights as a research subject.

The experimental procedure will be carried out in the University of Kentucky A.B. Chandler Hospital.

Direct measurements of the airway mucosal temperature will be performed before and at ten minutes after the SBP-Ag challenge. This miniature probe will be positioned in the airway lumen using an Olympus fiberoptic bronchoscope (model MP160F), and connected via a cable to a battery-operated thermometer (model FLL) manufactured also by Physitemp Instrument Inc. The probe (outside diameter of 0.4 mm) will be passed through the instrument channel (inner diameter: 2.0 mm) of the bronchoscope. By maneuvering the control knob of the bronchoscope, the blunted tip of the probe will be gently pressed against the airway mucosa at 5-6 different positions in segmental and sub-segmental bronchi, each for five to ten seconds. The entire protocol of the temperature measurement will require no more than 5 minutes to complete. The contact of the temperature probe on the airway mucosa should not cause any tissue damage, and is relatively non-invasive compared to other procedures involved in the routine bronchoscopy such as biopsy, cytology brushing, etc

Physical Examination: It will include assessment of subject's general condition, head and neck, chest and respiratory auscultation, cardiac auscultation, and limited abdominal, extremity and neurological exams.

Vital signs: Heart rate, blood pressure, body temperature and arterial oxygen saturation.

Screening Visits 1 and 2: Following procedures will occur on the screening visit after obtaining written informed consent.

* Collection of demographic information (Demographic data to be collected on screening visit will include name, initials, address, social security number, coded study number, medical record number, height, weight, age, race, ethnicity, gender, telephone number and email address.)
* Collection of medical and medication history
* Urine pregnancy test
* Vital signs
* Skin prick test
* Spirometry
* Limited physical examination
* Study eligibility review
* Whole lung allergen inhalation challenge
* Adverse Event assessment
* Concomitant medication

Visit 3 (Test Day 1)

* Review eligibility criteria
* Vital signs
* Spirometry
* Urine pregnancy test
* Physical examination
* Bronchoscopy with lavage
* Segmental allergen challenge
* Adverse Event assessment
* Concomitant medication

Visit 4 (Test Day 2)

* Review eligibility criteria
* Vital signs
* Spirometry
* Physical examination
* Bronchoscopy with lavage
* Adverse Event assessment
* Concomitant medication

Follow-up Phone Call. A follow-up phone call will take place 1 day following the last study visit. During this phone call the participant will be asked questions regarding any adverse events they may have experienced since the last visit along with the use of any concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* Diagnosis of well-controlled airway allergy with mild-intermittent asthma (a stable clinical condition with good asthma control) and demonstrating an allergen-specific airway response to inhaled allergen provocation.
* Pre-albuterol forced expiratory volume in the first second (FEV1) of >70% of the predicted value.
* Skin test positive to house dust mite, ragweed or cat hair.
* At least a 20% decrease in FEV1 during the immediate response following inhaled antigen challenge.
* Competent to understand and willing to grant written informed consent.

Exclusion Criteria:

* Inability to perform pulmonary function testing.
* History of any lung disease or disorder other than asthma.
* Major health problems such as autoimmune disease, heart disease, coronary artery disease, type I or type II diabetes, or uncontrolled hypertension.
* Pre-existing chronic infectious disease.
* Medication that is taken for other than for asthma, allergies or contraception.
* Inhaled corticosteroids or oral corticosteroids within 1 month of screening.
* Upper and lower respiratory infection within 1 month of screening.
* Unstable asthma as indicated by self report of increased symptoms or increased beta-agonist use over the 2 weeks preceding the screening visit.
* Pregnant or lactating females.
* History of smoking.
* History of noncompliance with medical regiments or subjects who are considered unreliable.
* Use of anti-platelet (i.e., aspirin, clopidogrel, etc) or anti-coagulant(coumadin, heparin, Xarelto®, etc) medication 5 days prior to bronchoscopy.

It is required that the subjects undergoing bronchoscopy are not on any anti-platelets (such as aspirin, clopidogrel, etc.) or anticoagulants (such as coumadin, heparin, Xarelto®, etc.) at least 5 days prior to the bronchoscopy. As such, subjects receiving any of these medications will be excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Airway tissue temperature | Immediately during experimental procedure (up to 10 minutes)
  Direct measurements of the airway mucosal temperature will be performed before and at ten minutes after the SBP-Ag challenge. By maneuvering the control knob of the bronchoscope, the blunted tip of the probe will be gently pressed against the airway mucosa at 5-6 different positions in segmental and sub-segmental bronchi, each for five to ten seconds. The entire protocol of the temperature measurement will require no more than 5 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Yuan Lee, PhD, Principal Investigator — University of Kentucky; Mehdi Khosravi, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Center for Clinical and Translational Science, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No